CLINICAL TRIAL: NCT06006650
Title: Pembrolizumab Plus Albumin Paclitaxel or 5-fluorouracil and Cisplatin Versus 5-fluorouracil and Cisplatin in Neoadjuvant Therapy for Resectable Esophageal Squamous Cell Carcinoma: a Prospective, Randomized Controlled Trial Study
Brief Title: Neoadjuvant Therapy for Stage II-IVA Resectable Esophageal Squamous Cell
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, yanxiaolong, Department of Thoracic Surgery at Tangdu Hospital, Air Force Medical University, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K202208-28
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Neoadjuvent; PD-1 Inhibitor; Chemotherapy; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab; Fluorouracil; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab Plus Albumin Paclitaxel and Cisplatin (Experimental): Preoperative neoadjuvant (pembrolizumab 200mg, d1 intravenously, q3w+ albumin paclitaxel 100mg/m2, d1/d8/d15 intravenously, q3w+ cisplatin 75mg/m2, d1 intravenously, q3w) 3 cycles + surgery + 16 cycles of postoperative pembrolizumab adjuvant therapy
  Interventions: Drug: Pembrolizumab, Albumin Paclitaxel, 5-fluorouracil, Cisplatin
- Pembrolizumab Plus 5-fluorouracil and Cisplatin (Active Comparator): Preoperative neoadjuvant (pembrolizumab 200mg, d1 intravenously, q3w+ 5-fluorouracil 800mg/m2, d1-5 intravenously, q3w+ cisplatin 75mg/m2, d1 intravenously, q3w) 3 cycles + surgery + 16 cycles of postoperative pembrolizumab adjuvant therapy
  Interventions: Drug: Pembrolizumab, Albumin Paclitaxel, 5-fluorouracil, Cisplatin
- 5-fluorouracil and Cisplatin (Active Comparator): Preoperative neoadjuvant (5-fluorouracil 800mg/m2, d1-5 intravenously, q3w+ cisplatin 75mg/m2, d1 intravenously, q3w) 3 cycles + surgery + 16 cycles of postoperative pembrolizumab adjuvant therapy
  Interventions: Drug: Pembrolizumab, Albumin Paclitaxel, 5-fluorouracil, Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab, Albumin Paclitaxel, 5-fluorouracil, Cisplatin — Pembrolizumab, Albumin Paclitaxel, 5-fluorouracil, Cisplatin

SUMMARY:
The aim of this study was to investigate the efficacy and safety of pembrolizumab combined with albumin paclitaxel and cisplatin versus albumin paclitaxel and cisplatin or 5-fluorouracil and cisplatin in neoadjuvant therapy for stage II-IVa resectable esophageal squamous cell carcinoma. The study plans to enroll 114 eligible patients who will be randomly assigned in a 1:1:1 ratio to receive 3 cycles of neoadjuvant immunochemotherapy (pembrolizumab plus albumin paclitaxel and cisplatin;Pembrolizumab plus 5-fluorouracil and cisplatin) or chemotherapy alone (5-fluorouracil and cisplatin), followed by surgery 3 weeks later, followed by 16 cycles of adjuvant immunotherapy (pembrolizumab).Patients were followed up for efficacy and safety during treatment.Tumor evaluation will be performed at screening, after neoadjuvant therapy, before surgery, and after adjuvant therapy until objective disease progression is confirmed.

DETAILED DESCRIPTION:
The aim of this study was to investigate the efficacy and safety of pembrolizumab combined with albumin paclitaxel and cisplatin versus albumin paclitaxel and cisplatin or 5-fluorouracil and cisplatin in neoadjuvant therapy for stage II-IVa resectable esophageal squamous cell carcinoma. The study plans to enroll 114 eligible patients who will be randomly assigned in a 1:1:1 ratio to receive 3 cycles of neoadjuvant immunochemotherapy (pembrolizumab plus albumin paclitaxel and cisplatin;Pembrolizumab plus 5-fluorouracil and cisplatin) or chemotherapy alone (5-fluorouracil and cisplatin), followed by surgery 3 weeks later, followed by 16 cycles of adjuvant immunotherapy (pembrolizumab).Patients were followed up for efficacy and safety during treatment.Tumor evaluation will be performed at screening, after neoadjuvant therapy, before surgery, and after adjuvant therapy until objective disease progression is confirmed.

Study Endpoints Primary Endpoints PCR: This was assessed by examining the postoperative pathological tissue for the absence of tumor cells in the primary tumor and lymph nodes.

Safety: Adverse reactions during neoadjuvant therapy were recorded following CTCAE version 5.0 guidelines. Perioperative complications were assessed using the Clavien-Dindo classification. Grade I complications included any deviation from the normal postoperative recovery process without requiring medical, surgical, endoscopic, or radiological intervention. Acceptable medical management included antiemetics, antipyretics, analgesics, diuretics, electrolytes, and physical therapy. Bedside open incisional infections were included under this category. Grade II complications were those that required medications beyond those used for treating Grade 1 complications, including blood transfusions and total parenteral nutrition. Grade III complications were those that required surgical, endoscopic, or radiological intervention. Grade IV complications were those considered life-threatening and requiring mid-term care or admission to an intensive care unit (including central nervous system complications, such as cerebral hemorrhage, ischemic stroke, and subarachnoid hemorrhage, and excluding transient ischemic attacks). Grade V complications included patient deaths.

Secondary Endpoints

1) Major pathological response (MPR) refers to the proportion of residual tumor cells in the primary tumor and lymph nodes in the postoperative pathological tissue being <10%, or the primary tumor completely disappearing, and the number of positive lymph nodes being ≤1. 2) R0 resection rate: R0 resection was defined as achieving negative upper and lower resection margins. 3) RECIST Criteria Assessment: Complete response (CR): complete response of target lesions; PR: >30% regression of target lesions; Non-CR/Non-PD: target lesions did not completely disappear and did not increase by >20%, or other new lesions appeared in the body; Stable disease (SD): target lesions were reduced or increased by <20%; Progressive disease (PD): target lesions had increased by >20%.

Statistical Methods The sample size was determined using Simon's two-stage design. With a minimum expected pCR of 20% and an expected pCR of 40%, a Type I error (α) of 0.05, and a Type II error of 80%, a sample size of 34 was calculated. In the first stage, 17 patients were enrolled. The study was carefully monitored to limit the number of pCR cases to three or below, and any increase in the risk of surgery and mortality due to the treatment regimen would have led to its discontinuation. All continuous variables were presented as frequencies. Statistical significance was set at P <0.05.

ELIGIBILITY:
Inclusion Criteria:

1.Pathological diagnosis: esophageal squamous cell carcinoma. 2.18-75 years old; 3.Clinical stage II-IVa; 4.no prior antitumor therapy, such as immunotherapy or chemoradiotherapy; 5.ECOG PS score 0-1. 6.Organs function well:Hemoglobin ≥100g/L, white blood cell count ≥4*10^9/L or neutrophil count ≥2.5*10^9/L, platelet count ≥100*10^9/L, serum total bilirubin level ≤1.5 times the upper limit of normal, aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal,Alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal, serum creatinine level below the upper limit of normal or creatinine clearance rate ≥60ml/min, urea nitrogen ≤200mg/L, urinary protein <+, if urinary protein +, 24-hour total protein must be <500mg, blood glucose:In patients with normal-range and/or diabetes under treatment but stable glycemic control, pulmonary function: baseline FEV1 of at least 2L;If the baseline FEV1 was <2L, the predicted FEV1 after surgery was >800ml, and the cardiac function was: no myocardial infarction within 1 year;Unstable angina pectoris;Asymptomatic severe arrhythmias;The centerless function is incomplete; 7.Non-surgically sterilized women, or women of reproductive age, need to use a medically approved contraceptive method (such as an intrauterine device, birth control pill, or condom) during and for 3 months after the end of the study treatment period.Women of childbearing age who were not surgically sterilized had to have a negative serum or urine HCG test within 72 hours before study enrollment.And must be non-lactation period;For male patients with partners of women of childbearing age, effective methods of contraception should be used during the trial period and within 3 months after the last dose of treatment; 8.Sign an informed consent form.

Exclusion Criteria:

1. Pathological findings suggest compound squamous cell carcinoma, including squamous adenocarcinoma, squamous cell carcinoma, carcinosarcoma, sarcomatoid carcinoma, etc.
2. History of subtotal gastrectomy;
3. accompanied by a second primary cancer;
4. Tumor metabolic imaging prior to treatment suggested distant metastasis.
5. people who have previously received chemoradiotherapy;
6. preesophageal perforation signs
7. pregnant women of reproductive age;
8. Any active autoimmune disease or a history of autoimmune disease (such as autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, etc.);
9. People with the following active infectious diseases, including active tuberculosis, hepatitis, and known human immunodeficiency virus (HIV) infection;
10. Someone who has a known or concomitant hemorrhagic disease or other uncontrollable disease that cannot be treated surgically;
11. Physical examination or clinical trial findings that researchers believe could interfere with the outcome or put the patient at increased risk of treatment complications;
12. A previous history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis requiring hormone therapy, or any clinically documented active interstitial lung disease, and the presence of idiopathic pulmonary fibrosis on CT scan at baseline;Uncontrolled massive pleural or pericardial effusion;
13. unstable systemic diseases (active infection, moderately severe chronic obstructive pulmonary disease (copd), poorly controlled hypertension, unstable angina and congestive heart failure, 6 months occurrence of myocardial infarction, drug control severe mental disorders, liver, kidney or other metabolic disease, nerve mental disease such as Alzheimer 's disease);
14. Gastrointestinal dysfunction, malabsorption syndrome, active gastrointestinal ulcers;
15. Previously treated with anti-PD-1 or anti-PD-L1 antibodies;
16. Receiving any investigational drug within 4 weeks before the first use of the investigational drug;
17. Enroll in another clinical study at the same time, unless it's an observational (non-intervention) clinical study or an intervention clinical study follow-up;
18. Subjects who require systematic treatment with corticosteroids (equivalent dose of prednisone > 10 mg per day) or other immunosuppressive agents within 2 weeks prior to the first use of the study drug, except for the use of corticosteroids for local esophageal inflammation and prevention of allergy, nausea, and vomiting.Other special circumstances, need to communicate with the sponsor.In the absence of active autoimmune disease, inhaled or topical steroids and adrenocorticosteroid replacement at doses > 10mg/ day in response to prednisone are permitted;
19. People who have been vaccinated with anti-tumor vaccine or who have been vaccinated with live vaccine within 4 weeks prior to the first administration of the study drug;
20. Major surgery or severe trauma within 4 weeks before the first use of the study drug;
21. Congenital or acquired immunodeficiency disease or a history of organ transplantation;A history of allergies to monoclonal antibodies, albumin paclitaxel, 5-fluorouracil, cisplatin, and other platinum-based drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) | up to 4 months
  Pathologic complete response rate (pCR)

SECONDARY OUTCOMES:
Major pathological response(MPR) | up to 4 months
  Major pathological response(MPR)
Event free survival(EFS) | up to 10 years
  Event free survival(EFS)
Overall survival(OS) | up to 10 years
  Overall survival(OS)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Yan, MD, Principal Investigator — Tang-Du Hospital
Locations (3):
- China (3):
  - Tangdu Hospital of the Fourth Millitary Medical University, Xi'an, Shaanxi
  - Hongtao Duan, Xi’an, Shanxi
  - Tangdu Hospital, the Air Force Military University, Xi'an

IPD SHARING:
Plan to Share IPD: No